CLINICAL TRIAL: NCT03030001
Title: PD-1 Antibody Expressing Chimeric Antigen Receptor T Cells for Mesothelin Positive Advanced Malignancies
Brief Title: PD-1 Antibody Expressing CAR T Cells for Mesothelin Positive Advanced Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ningbo Cancer Hospital (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2017-01-P01
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Solid Tumor, Adult; Advanced Cancer
Keywords: mesothelin; PD-1; CAR T; solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody expressing CAR-T cells (Experimental): PD-1 antibody expressing mesothelin specific CAR-T cells
  Interventions: Biological: PD-1 antibody expressing mesothelin specific CAR-T cells

INTERVENTIONS:
Biological: PD-1 antibody expressing mesothelin specific CAR-T cells — Patients will receive an IV infusion of PD-1 antibody expressing mesothelin specific CAR engineered peripheral blood leukocyte. On day 21, cells will be infused intravenously (i.v.) on the Patient Care Unit over 20 to 30 minutes.

SUMMARY:
This is a single-arm, open-label, one center, dose escalation clinical study, to determine the safety and efficacy of infusion of autologous T cells engineered to express immune checkpoint antibody and chimeric antigen receptor targeting mesothelin in adult patients with mesothelin positive, recurrent or refractory malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Relapsed or refractory advanced solid malignancies.
* 2. Progressive disease and no response to current therapy.
* 3. Patients must have previously received at least one standard therapy for their cancer (if available) and have been either non-responders (progressive disease) or have recurred. And patients are willing to attend the clinical trial.
* 4. Gender unlimited, age from 18 years to 80 years.
* 5. Life expectancy≥6 months.
* 6. ECOG (Eastern Cooperative Oncology Group) performance status of 0-2.
* 7. Adequate venous access for apheresis, and no other contraindications for leukapheresis ; Peripheral venous access ；no contraindication of lymphocyte separation.
* 8. IHC( immuno-histochemistry) result of tumor tissue： mesothelin positive for ：frequency≥2，intensity≥2 +. The percentage of tumor cell nuclei stained (0, no staining; 1, ≤10%; 2, 10-50% and 3, >50%) and the staining intensity (ranging from 0 to 3+).
* 9. Adequate hepatic function, renal function and bone marrow function：WBC≥3.0×109/L,PLT≥60×109/L,HGB≥85g/L,LY≥0.7×109/L; Alanine aminotransferase/Aspartate transaminase(ALT/AST) 2.5 times the upper limit of the normal value, total bilirubin(TBiL) 1times the upper limit of the normal value, Serum creatinine1.5 times the upper limit of the normal value.
* 10. Willing and able to understand and sign the Informed Consent Document.
* 11. Women of child-bearing age must have evidence of negative pregnancy test. Patients must be willing to practice birth control during and for four months following treatment.

Exclusion Criteria:

* 1. Life expectancy6 months.
* 2. Patients with uncontrolled active infection will be excluded.
* 3. Patients with severe heart and lung dysfunction; uncontrolled hypertension, unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> New York Heart Association Class II), or myocardial infarction within 6 months of study will be excluded; aberrant pulmonary function testing: with a forced expiratory volume (FEV) of <30%(predicted), diffusion capacity of the lung for carbon monoxide (DLCO) (corrected) <30% and oxyhemoglobin saturation90% will be excluded.
* 4. Patients with severe liver and kidney dysfunction or chronic diseases of important organs will be excluded.
* 5. Patients with active autoimmune disease requiring immunosuppressive therapy will be excluded.
* 6. Patients requiring corticosteroids (other than inhaled) will be excluded.
* 7. Patients with other severe diseases or situations improper for the research will be excluded, including neurologic disease, mental disease, immune disease, metabolic disease, and contagious disease.
* 8. Pregnant and/or lactating women will be excluded.
* 9. Patients who have had other bio-therapy in the past 4 weeks.
* 10. Patients who are participating or participated any other clinical trials in latest 30 days will be excluded.
* 11. Patients with the subject suffering disease affects the understanding of informed consent or complying with study protocol will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-15 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion of autologous mesothelin specific CAR T cells | 2 years
  Safety of infusion of autologous mesothelin specific CAR T cells with PD-1 antibody expressing in patients with relapsed or refractory advanced solid malignancies using the NCI CTCAE V4.0 criteria

SECONDARY OUTCOMES:
the response evaluation criteria of solid tumor | 2 years
  Defined as the overall response rate (ORR), the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) based on the response evaluation criteria in solid tumor version 1.1 (RECIST1.1).
progression free survival | 1 year
overall survival | 2 years

OTHER OUTCOMES:
Change of life quality after treatment | 2 years
proliferation and persistence of mesothelin specific CAR T cells in patients after treatment | 6 months
expression of PD-1 antibody in patients after treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Qijun Qian, PhD, Study Chair — Shanghai Cell Therapy Engineering Research Institute
Locations (1):
- Ningbo No.5 Hospital (Ningbo Cancer Hospital), Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided